CLINICAL TRIAL: NCT00770445
Title: Impact of Pioglitazone, Metformin and the Combination of Both on Cardiovascular Risk in Insulin-treated Patients With Type 2 Diabetes - The PIOcomb Study
Brief Title: Efficacy of Pioglitazone and Metformin on Cardiovascular Risk in Subjects With Insulin-Treated Type 2 Diabetes Mellitus.
Acronym: PIOcomb
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Pharma GmbH, Aachen (Germany)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATS K028; 2007-006706-14 (EudraCT Number); DE-PIO-028 (Other: Takeda ID); U1111-1113-1888 (Registry Identifier: WHO)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone; Insulin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pioglitazone 15mg BID (Experimental): Insulin therapy added
  Interventions: Drug: Pioglitazone and insulin
- Pioglitazone 15mg + Metformin 850mg BID (Experimental): Insulin Therapy Added
  Interventions: Drug: Pioglitazone and metformin and insulin
- Metformin 850mg BID (Active Comparator): Insulin therapy added
  Interventions: Drug: Metformin and insulin

INTERVENTIONS:
Drug: Pioglitazone and insulin — Pioglitazone 15 mg, tablets, orally, twice daily and metformin placebo-matching tablets, orally, twice daily and insulin glargine stable dose for up to 24 weeks.
  Other Names: ACTOS®
  Arms: Pioglitazone 15mg BID
Drug: Pioglitazone and metformin and insulin — Pioglitazone 15 mg, tablets, orally, twice daily and metformin 850 mg, tablets, orally, twice daily and insulin glargine stable dose for up to 24 weeks.
  Other Names: ACTOS®
  Arms: Pioglitazone 15mg + Metformin 850mg BID
Drug: Metformin and insulin — Pioglitazone placebo-matching tablets, orally, twice daily and metformin 850 mg, tablets, orally, twice daily and insulin glargine stable dose for up to 24 weeks.
  Arms: Metformin 850mg BID

SUMMARY:
The purpose of this study is to determine the Anti-Inflammation Effects of Pioglitazone, twice daily (BID), and Pioglitazone/Metformin Combination Therapy BID in Type 2 Diabetes Subjects Treated with Insulin.

DETAILED DESCRIPTION:
It is established that matrix metalloproteinases play an essential role in the degradation of collagen and other extra cellular matrix macromolecules. In addition, matrix metalloproteinases are implicated in plaque rupture through their capacity to thin the protective cap of the plaque, thus rendering it more vulnerable. In fact, matrix metalloproteinase-9 levels are elevated in patients with unstable plaques and in patients with acute coronary syndrome. In patients with type 2 diabetes mellitus, matrix metalloproteinase-1 and matrix metalloproteinase-9 levels are usually elevated and the atherosclerotic plaques are more vulnerable compared to non-diabetic patients, confirming the role of this proteinase in the development of acute coronary syndrome. Therefore, therapeutic strategies that reduce blood glucose levels and attenuate inflammation and matrix metalloproteinases activity may be a tool for reducing cardiovascular risk in patients with diabetes.

The purpose of this trial is to investigate whether the anti-inflammatory effects of pioglitazone are maintained and sustained over a longer observation period when given in combination with insulin in comparison to the metformin plus insulin combination. The duration of treatment for patients completing the study is approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Has Diabetes Mellitus type 2.
* A glycosylated hemoglobin level greater than or equal to 6.5% and less than 8.5%.
* Treatment with the following insulins with or without Oral Antidiabetic Therapy since 3 months:

  * Long acting basal insulin analogs
  * NPH insulin
  * Combination insulin with 1-2 daily doses except intensified insulin therapies.
* A body mass index greater than or equal to 25.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* Has a history of type 1 diabetes mellitus.
* Has uncontrolled hypertension (systolic blood pressure greater than 160mmHg and/or diastolic blood pressure greater than 95mmHg) or change of antihypertensive treatment within the last 2 weeks.
* Has acute infections.
* Has anamnestic history of hypersensitivity to the study drugs or to drugs with similar chemical structure.
* Has a history of severe or multiple allergies.
* History of drug or alcohol abuse in the past 5 years
* A history of significant cardiovascular (New York Heart Association stage I - IV), respiratory, gastrointestinal, hepatic (Alanine Aminotransferase and/or Aspartate Aminotransferase greater than 2.5 times the upper limit of the normal reference range), renal (serum creatinine greater than 1.2 mg/dL in women and greater than 1.5 mg/dL in men, Glomerular Filtration Rate less than 60 ml/min as estimated by the Cockroft-Gault formula), neurological, psychiatric and/or hematological disease as judged by the investigator
* History of macular edema.
* State after kidney transplantation.
* Serum potassium greater than 5.5 mmol/L.
* History of primary hyperaldosteronism.
* Acute myocardial infarction, open heart surgery or cerebral event (stroke/ Transitory Ischemic Attack) within the previous 12 months.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Pre-treatment with gemfibrozil within the last 12 weeks.
  * Pre-treatment with rifampicin within the last 12 weeks.
  * Treatment with thiazolidinediones within the past 3 months.
  * If statin therapy applicable: Change of medication within the last 4 weeks.
  * Has used non-steroidal anti-inflammatory agents including low dose ASA or Cox-2-inhibitors if therapy has been initiated within the last 4 weeks.
  * Treatment with any other investigational drug within 4 weeks before trial entry.
* Any elective surgery during study participation.
* Have had more than one unexplained episode of severe hypoglycemia (defined as requiring assistance of another person due to disabling hypoglycemia) within 6 months prior to screening visit.
* History of dehydration, precoma diabeticorum or shock or diabetic ketoacidosis within the past year prior to screening visit.
* Acute or scheduled investigation with iodine containing radiopaque material.
* Uncontrolled unstable angina pectoris.
* Medical history of acute and clinically relevant pericarditis, myocarditis, endocarditis, recent pulmonary embolism, hemodynamic relevant aortic stenosis, aortic aneurysm.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Matrix Metallo Proteinase 9. | Baseline and Week 24.
  The change between Matrix Metallo Proteinase 9 collected at final visit or week 24 and Matrix Metallo Proteinase 9 collected at baseline.

SECONDARY OUTCOMES:
Change from Baseline in 24-hour Blood Pressure Profile. | Baseline and Week 24.
  The change between the 24-hour Blood Pressure Profile recorded at final visit or week 24 and 24-hour Blood Pressure Profile recorded at baseline.
Change from Baseline in Intima Media Thickness. | Baseline and Week 24.
  The change between the value of Intima Media Thickness measured at final visit or week 24 and Intima Media Thickness measured at baseline.
Change from Baseline in 24-hour Urinary Sample. | Baseline and Week 24.
  The change between the value of urine participants collect 24 hours before final visit or week 24 and urine participants collect 24 hours before baseline.
Change from Baseline in N-terminal Pro-hormone Brain Natriuretic Peptide. | Baseline and Week 24.
  The change between the value of N-terminal Pro-hormone Brain Natriuretic Peptide collected at final visit or week 24 and N-terminal Pro-hormone Brain Natriuretic Peptide collected at baseline.
Change from Baseline in 8-iso Prostaglandin F2 alpha. | Baseline and Week 24.
  The change between the value of 8-iso Prostaglandin F2 alpha collected at final visit or week 24 and 8-iso Prostaglandin F2 alpha collected at baseline.
Change from Baseline in Albumin. | Baseline and Week 24.
  The change between the value of Albumin collected at final visit or week 24 and Albumin collected at baseline.
Change from Baseline in Creatinine. | Baseline and Week 24.
  The change between the value of Creatinine collected at final visit or week 24 and Creatinine collected at baseline.
Change from Baseline in C/A-quotient. | Baseline and Week 24.
  The change between the value of C/A-quotient collected at final visit or week 24 and C/A-quotient collected at baseline.
Change from Baseline in Homeostasis Model Assessment - Insulin Sensitivity. | Baseline and Week 24.
  The change between Homeostasis Model Assessment of Insulin Sensitivity collected at final visit or week 24 and Homeostasis Model Assessment of Insulin Sensitivity collected at baseline. Homeostatis Model Assessment measures insulin sensitivity, calculated by fasting insulin times fasting glucose, divided by a constant (22.5).
Change from Baseline in Total Cholesterol. | Baseline and Week 24.
  The change between the value of Total Cholesterol collected at final visit or week 24 and Total Cholesterol collected at baseline.
Change from Baseline in Low-Density Lipoprotein. | Baseline and Week 24.
  The change between the value of Low-Density Lipoprotein collected at final visit or week 24 and Low-Density Lipoprotein collected at baseline.
Change from Baseline in High-Density Lipoprotein. | Baseline and Week 24.
  The change between the value of High-Density Lipoprotein collected at final visit or week 24 and High-Density Lipoprotein collected at baseline.
Change from Baseline in Triglycerides. | Baseline and Week 24.
  The change between the value of Triglycerides collected at final visit or week 24 and Triglycerides collected at baseline.
Change from Baseline in Glycosylated Hemoglobin. | Baseline and Week 24.
  The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at final visit or week 24 and Glycosylated Hemoglobin collected at baseline.
Change from Baseline in Glucose. | Baseline and Week 24.
  The change between the value of Glucose collected at final visit or week 24 and Glucose collected at baseline.
Change from Baseline in Insulin. | Baseline and Week 24.
  The change between the value of Insulin collected at final visit or week 24 and Insulin collected at baseline.
Change from Baseline in Intact Proinsulin. | Baseline and Week 24.
  The change between the value of Intact Proinsulin collected at final visit or week 24 and Intact Proinsulin collected at baseline.
Change from Baseline in C-peptide. | Baseline and Week 24.
  The change between the value of C-peptide collected at final visit or week 24 and C-peptide collected at baseline.
Change from Baseline in Adiponectin. | Baseline and Week 24.
  The change between the value of Adiponectin collected at final visit or week 24 and Adiponectin collected at baseline.
Change from Baseline in High Molecular Weight Adiponectin. | Baseline and Week 24.
  The change between the value of High Molecular Weight Adiponectin collected at final visit or week 24 and High Molecular Weight Adiponectin collected at baseline.
Change from Baseline in High-Sensitivity C-Reactive Protein. | Baseline and Week 24.
  The change between the value of High-Sensitivity C-Reactive Protein collected at final visit or week 24 and High-Sensitivity C-Reactive Protein collected at baseline.
Change from Baseline in Fibrinogen. | Baseline and Week 24.
  The change between the value of Fibrinogen collected at final visit or week 24 and Fibrinogen collected at baseline.
Change from Baseline in E-selectin | Baseline and Week 24.
  The change between the value of E-selectin collected at final visit or week 24 and E-selectin collected at baseline.
Change from Baseline in Nuclear Factor-kappa B. | Baseline and Week 24.
  The change between the value of Nuclear Factor-kappa B collected at final visit or week 24 and Nuclear Factor-kappa B collected at baseline.
Change from Baseline in Plasminogen Activator Inhibitor-1. | Baseline and Week 24.
  The change between the value of Plasminogen Activator Inhibitor-1 collected at final visit or week 24 and Plasminogen Activator Inhibitor-1 collected at baseline.
Change from Baseline in Nitrotyrosine. | Baseline and Week 24.
  The change between the value of Nitrotyrosine collected at final visit or week 24 and Nitrotyrosine collected at baseline.
Change from baseline in Insulin Consumption. | Baseline and Week 24.
  The change between the value of Insulin collected at final visit or week 24 and Insulin collected at baseline.
Change from Baseline in Endothelial Function measured by Laser-Doppler-flowmetry. | Baseline and Week 24.
  The change between the value of Endothelial Function measured at final visit or week 24 and Endothelial Function measured at baseline.
Change from Baseline in Body Weight. | Baseline and Week 24.
  The change between the value of the participant's Body Weight recorded at final visit or week 24 and the participant's Body Weight recorded at baseline.
Change from Baseline in Electrocardiograms | Baseline and Week 24.
  The change between the value of Electrocardiograms measured at final visit or week 24 and Electrocardiograms measured at baseline.
Change from Baseline in Alanine Aminotransferase Laboratory Safety Variable. | Baseline and Week 24.
  The change between the value of Alanine Aminotransferase collected at final visit or week 24 and Alanine Aminotransferase collected at baseline.
Change from Baseline in Aspartate Aminotransferase Laboratory Safety Variable. | Baseline and Week 24.
  The change between the value of Aspartate Aminotransferase collected at final visit or week 24 and Aspartate Aminotransferase collected at baseline.
Change from Baseline in Gamma-glutamyl transferase Laboratory Safety Variable. | Baseline and Week 24.
  The change between the value of Gamma-glutamyl transferase collected at final visit or week 24 and Gamma-glutamyl transferase collected at baseline.
Change from Baseline in Glomerular Filtration Rate Laboratory Safety Variable. | Baseline and Week 24.
  The change between the value of Glomerular Filtration Rate collected at final visit or week 24 and Glomerular Filtration Rate collected at baseline.
Change from Baseline in Alkaline Phosphatase Laboratory Safety Variable. | Baseline and Week 24.
  The change between the value of Alkaline Phosphatase collected at final visit or week 24 and Alkaline Phosphatase collected at baseline.
Change from Baseline in Leucocytes Laboratory Safety Variable. | Baseline and Week 24.
  The change between the value of Leucocytes collected at final visit or week 24 and Leucocytes collected at baseline.
Change from Baseline in Hemoglobin Laboratory Safety Variable. | Baseline and Week 24.
  The change between the value of Hemoglobin collected at final visit or week 24 and Hemoglobin collected at baseline.
Change from Baseline in Thrombocytes Laboratory Safety Variable. | Baseline and Week 24.
  The change between the value of Thrombocytes collected at final visit or week 24 and Thrombocytes collected at baseline.
Change from Baseline in Creatinine Kinase Laboratory Safety Variable. | Baseline and Week 24.
  The change between the value of Creatinine Kinase collected at final visit or week 24 and Creatinine Kinase collected at baseline.
Change from Baseline in Creatinine Laboratory Safety Variable. | Baseline and Week 24.
  The change between the value of Creatinine collected at final visit or week 24 and Creatinine collected at baseline.
Change from Baseline in Capillary Blood Glucose Laboratory Safety Variable. | Baseline and Week 24.
  The change between the value of Capillary Blood Glucose collected at final visit or week 24 and Capillary Blood Glucose collected at baseline.
Change from Baseline in Potassium Laboratory Safety Variable. | Baseline and Week 24.
  The change between the value of Potassium collected at final visit or week 24 and Potassium collected at baseline.
Change from Baseline in Circadian (7 point) Blood Glucose Profile (Week 24). | Baseline and Week 24.
  The change between Circadian Blood Glucose measured before week 24 or final visit and Circadian Blood Glucose measured before baseline. Participants measure their blood glucose levels 7 times (before and after breakfast, before and after lunch, before and after dinner and before going to bed) on two arbitrary days and record these measurements in their diaries.
Change from Baseline in Circadian (7 point) Blood Glucose Profile (Week 12). | Baseline and Week 12.
  The change between Circadian Blood Glucose measured before week 12 and Circadian Blood Glucose measured before baseline. Participants measure their blood glucose levels 7 times (before and after breakfast, before and after lunch, before and after dinner and before going to bed) on two arbitrary days and record these measurements in their diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda Pharma GmbH, Aachen (Germany)
Locations (18):
- Germany (18):
  - Lichtenfels, Bavaria
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Kassel, Hesse
  - Wiesbaden, Hesse
  - Bad Oeynhausen, North Rhine-Westphalia
  - Dinslaken, North Rhine-Westphalia
  - Duisburg, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Diez, Rhineland-Palatinate
  - Landau, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Leipzig, Saxony
  - Berlin, State of Berlin
  - Jena, Thuringia

REFERENCES:
- See also: ACTOSPLUS MET® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOPLUSMETPI